CLINICAL TRIAL: NCT06905392
Title: AQT90 FLEX NTproBNP2 Test Kit Matrix Comparison and Sample Stability Verification Study
Status: Recruiting | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-087459
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-08

CONDITIONS: Diagnostic Tests

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to establish the correlation between sample matrices, and to determine the sample stability for the NTproBNP2 Test Kit on the AQT90 FLEX analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to understand given information and demonstrate willingness and ability to voluntarily give a signed, valid written informed consent to participate in the study.
* Subjects must be 18 years of age or older.
* Subjects with expected NT-proBNP concentrations within the measuring range of NTproBNP2 Test Kit.

Exclusion Criteria:

* Subjects known to be pregnant or breast-feeding.
* Subjects previously enrolled in the study.
* Subject, who has withdrawn consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient population with expected NT-proBNP concentrations within the measuring range of NTproBNP2 Test Kit.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation | 5 month
  To establish a correlation between sample matrices
Stability | 5 month
  To determine sample stability with the NTproBNP2 Test Kit on the AQT90 FLEX analyzer

CONTACTS AND LOCATIONS:
Locations (5):
- Hennepin Healthcare (Research Institute/ Minneapolis Medical Research Foundation), Minneapolis, Minnesota, United States
- Spain (4):
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Clinica Universidad de Navarra, Pamplona
  - Hospital Clinico Universitario de Santiago Compostela, Santiago de Compostela
  - Servicio Andaluz de Salud (SAS) - Hospital San Juan de la Cruz, Ùbeda